CLINICAL TRIAL: NCT04394884
Title: Pathogenesis of BTK-mediated Hyper-Inflammatory Responses in COVID-19
Brief Title: Pathogenesis of BTK-mediated Hyper-Inflammatory Responses in COVID-19 (RESPOND)
Status: Withdrawn | Type: Observational
Why Stopped: Study never started, no subjects enrolled.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200114; 20-I-0114
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: Sample Collection; Immunological Mechanisms; SARS-CoV-2; Serelogic Response; Imflammatory Pathway
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- COVID-19 -: will receive BTK therapy for other reasons
- COVID-19 + BTK: will receive BTK therapy
- COVID-19 + No BTK: will not receive BTK therapy

SUMMARY:
Background:

Coronavirus disease 2019 (COVID-19) is an acute respiratory syndrome. It is caused by the SARS-CoV-2 virus. People with severe COVID-19 infection have a hyper-inflammatory response. Bruton tyrosine kinase (BTK) plays a role in the innate immune system. BTK inhibition can be used to target the innate immune system that appears to contribute to mortality. This could be an effective way to help the inflammatory responses in people with COVID-19.

Objective:

To learn more about the immunologic mechanisms by which BTK inhibition may decrease hyper-inflammatory responses in people with COVID-19.

Eligibility:

People ages 18 and older in one of the following groups:

* They are in the hospital with COVID-19. They will or will not be treated with a BTK inhibitor.
* They do not have COVID-19. They are or are not in the hospital. They will be treated with a BTK inhibitor for a reason other than COVID-19.

Design:

Participants will be screened with a review of their demographic and clinical information. Their medical history will be reviewed. If they have COVID-19, their symptoms will be assessed.

Participants will give 3-4 blood samples. These may be taken through a vein. They may also be taken through an existing central venous catheter.

Participants may give a stool sample. This will be collected by nursing staff. It will be collected using a stool collection vial. Stool collection is optional.

Participants samples will be collected over about 7 days. These will be used for research and genetic testing.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an acute respiratory syndrome caused by the novel coronavirus severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). Severe COVID-19 infection is associated with a hyper-inflammatory response and evidence of innate immune cell activation. Bruton tyrosine kinase (BTK) plays a central role in innate immune cell signaling and activation and BTK inhibition represents a promising therapeutic strategy for ameliorating excessive inflammatory responses in patients with COVID-19. Understanding the mechanisms by which BTK inhibition modulates the host inflammatory response in patients with COVID-19 is critical in order to better understand COVID-19 pathogenesis.

In this multisite natural history laboratory study, hospitalized patients with COVID-19 (n=80) will be recruited at Walter Reed National Military Medical Center and The Johns Hopkins Hospital. Forty of these patients will be recipients of BTK inhibition, either as part of their standard clinical care or in another clinical trial. The other 40 will not be recipients of BTK inhibition and will serve as a control group. A third group of patients without COVID-19 (n=40) who will be recipients of BTK inhibition for other clinical indications will also be enrolled as a second control group.

Participants will have three or four longitudinal blood draws and may be asked to provide stool samples. All specimens and data will be coded and sent to the National Institutes of Health (NIH) for research analysis. Only site investigators will have access to the code s key for their respective sites; the NIH investigators will not have the keys. Coded blood samples will be used for genetic testing, transcriptional analyses, deep immunological phenotyping, soluble biomarker analysis, and other research tests. Coded clinical and laboratory data from routine care (e.g., basic demographic information, vital signs, medications, clinical labs, and radiologic imaging findings) will also be captured. Coded stool samples may be collected as part of this study to determine whether viable SARS-CoV-2 is present in stool, which will help advance our understanding of pathogenesis and enteric transmission.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to provide informed consent, and
2. Men and women >=18 years of age at the time of signing the informed consent form, and
3. Diagnosis of COVID-19 in hospitalized patients with hypoxemia (SpO2 less than or equal to 94% on room air), with plan to receive or not receive BTK inhibition for clinical or for external research study purposes, or
4. Does not have COVID-19 and does have plan to receive BTK inhibition therapy for a clinical indication other than COVID-19 (either hospitalized or not).

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Documented history of hemoglobin from most recent blood draw <7g/dL if known.
2. Pregnant or breastfeeding.
3. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people admitted to the participating sites who have COVID-19 or some other disease were they are already receiving or will receive BTK therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
To characterize the immunologic mechanisms by which BTK inhibition may ameliorate hyper- inflammatory responses in patients with COVID-19. | day 0, 1,3,7
  Inflammatory pathway analyses following BTK inhibition in COVID-19 patients.

SECONDARY OUTCOMES:
1. Characterization of TLR3 and TLR7/8-dependent immunologic phenotypes in COVID-19 patients before and after BTK inhibition. | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.
2. Evaluation of mechanisms of immune cell-specific activation, cytokine production, exhaustion and apoptosis in COVID-19 patients before and after BTK inhibition. | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.
3. Transcriptional, chromatin, and epigenetic profiling of immune cells at the single cell level in COVID-19 patients before and after BTK inhibition. | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.
4. Longitudinal evaluation of TCR and BCR repertoire development in COVID-19 patients before and after BTK inhibition. | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.
5. Characterization of SARS- CoV-2 serological responses in COVID-19 patients with and without BTK inhibition. | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.
6. Characterization of genetic variants that correlate with disease severity and/or response to BTK inhibition treatment. | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.
7. Evaluation of soluble biomarkers as surrogate markers of hyper- inflammation/prognosis and of response to BTK inhibition therapy in COVID-19 patients | day 0, 1,3,7
  Transcriptomic, genomic, serological and immunologic analyses of response to BTK inhibition therapy in COVID- 19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michail S Lionakis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Walter Reed National Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0114.html